CLINICAL TRIAL: NCT05740774
Title: Feasibility of 3D Ultrasound in the Assessment of Resection Margins During Surgery for Squamous Cell Carcinoma of the Tongue: a Comparison With Histopathology
Brief Title: Surgical Margin Assessment by 3D Ultrasound
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Fatemeh Makouei, Biomedical Engineer, PhD, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21017915a
Record Dates: First submitted 2023-02-11; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Tongue Cancer; Squamous Cell Carcinoma; Head and Neck Cancer
Keywords: 3D ultrasound; Histopathology; Ultrasonography; Three dimensional imaging; cancer diagnosis; tongue tumor
MeSH Terms: conditions — Tongue Neoplasms; Carcinoma, Squamous Cell; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tongue tumor resection (Experimental)
  Interventions: Diagnostic Test: 3D ultrasound

INTERVENTIONS:
Diagnostic Test: 3D ultrasound — 3D ultrasound scanning of the resected tongue tumor will be performed. The margin analysis will be made using the 3D ultrasound image.

SUMMARY:
Complete removal of cancer encircled by a secure margin of healthy tissue is the aim of surgical oncology. A close or positive surgical margin reported by pathologist typically ends in adjuvant therapies (re-surgery and/or radiotherapy), which come with prognostic risks and financial cost. Therefore, ex-vivo imaging of removed cancer tissue may assist in margin evaluation. In this study, investigators aimed to investigate the correlation of 3D ultrasound to histopathology to assess tongue tumor margin status.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven oral tongue squamous cell carcinoma scheduled for surgical treatment
* T1-T2 staging on cross-sectional imaging

Exclusion Criteria:

* Age < 18 yrs
* T3-T4 staging
* Unable to understand the verbal or written information
* Prior radiotherapy treatment of oral cavity cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Correlation of the surgical margin measurements of the 3D ultrasound to histopathology | 2 weeks
  The smallest margin will be measured in mm on 3D ultrasound image of the ex-vivo surgical specimen. Correlation of the measurement to the final histopathology result will be investigated.
Diagnostic accuracy | 2 weeks
  number of margins correctly classified as free (> 5 mm), close (< 5 mm) or positive (<1 mm) margin

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, København Ø, Dk-015, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP
Time Frame: Available for 5 years

REFERENCES:
- [Background] Chinn SB, Myers JN. Oral Cavity Carcinoma: Current Management, Controversies, and Future Directions. J Clin Oncol. 2015 Oct 10;33(29):3269-76. doi: 10.1200/JCO.2015.61.2929. Epub 2015 Sep 8. PMID 26351335
- [Background] de Koning KJ, van Es RJJ, Klijn RJ, Breimer GE, Willem Dankbaar J, Braunius WW, van Cann EM, Dieleman FJ, Rijken JA, Tijink BM, de Bree R, Noorlag R. Application and accuracy of ultrasound-guided resections of tongue cancer. Oral Oncol. 2022 Oct;133:106023. doi: 10.1016/j.oraloncology.2022.106023. Epub 2022 Jul 25. PMID 35901543
- [Background] Tarabichi O, Bulbul MG, Kanumuri VV, Faquin WC, Juliano AF, Cunnane ME, Varvares MA. Utility of intraoral ultrasound in managing oral tongue squamous cell carcinoma: Systematic review. Laryngoscope. 2019 Mar;129(3):662-670. doi: 10.1002/lary.27403. Epub 2018 Aug 27. PMID 30151976
- [Background] Klein Nulent TJW, Noorlag R, Van Cann EM, Pameijer FA, Willems SM, Yesuratnam A, Rosenberg AJWP, de Bree R, van Es RJJ. Intraoral ultrasonography to measure tumor thickness of oral cancer: A systematic review and meta-analysis. Oral Oncol. 2018 Feb;77:29-36. doi: 10.1016/j.oraloncology.2017.12.007. Epub 2017 Dec 18. PMID 29362123
- [Background] Narayana HM, Panda NK, Mann SB, Katariya S, Vasishta RK. Ultrasound versus physical examination in staging carcinoma of the mobile tongue. J Laryngol Otol. 1996 Jan;110(1):43-7. doi: 10.1017/s0022215100132682. PMID 8745780
- [Background] Makouei F, Ewertsen C, Agander TK, Olesen MV, Pakkenberg B, Todsen T. 3D Ultrasound versus Computed Tomography for Tumor Volume Measurement Compared to Gross Pathology-A Pilot Study on an Animal Model. J Imaging. 2022 Dec 19;8(12):329. doi: 10.3390/jimaging8120329. PMID 36547494
- [Background] de Koning KJ, Koppes SA, de Bree R, Dankbaar JW, Willems SM, van Es RJJ, Noorlag R. Feasibility study of ultrasound-guided resection of tongue cancer with immediate specimen examination to improve margin control - Comparison with conventional treatment. Oral Oncol. 2021 May;116:105249. doi: 10.1016/j.oraloncology.2021.105249. Epub 2021 Mar 26. PMID 33774501
- [Background] Schmidt Jensen J, Jakobsen KK, Mirian C, Christensen JT, Schneider K, Nahavandipour A, Wingstrand VL, Wessel I, Tvedskov JF, Frisch T, Christensen A, Specht L, Andersen E, Lelkaitis G, Gronhoj C, von Buchwald C. The Copenhagen Oral Cavity Squamous Cell Carcinoma database: protocol and report on establishing a comprehensive oral cavity cancer database. Clin Epidemiol. 2019 Aug 19;11:733-741. doi: 10.2147/CLEP.S215399. eCollection 2019. PMID 31695503